CLINICAL TRIAL: NCT05159063
Title: Correlation of Internal Jugular and Inferior Vena Cava Diameter Variation on Bedside Ultrasound With Invasive Right Heart Catheterization
Brief Title: Bedside Ultrasound for Fluid Estimation
Status: Completed | Type: Observational
Sponsor: Gaurang Vaidya (Other)
Responsible Party: Sponsor-Investigator, Gaurang Vaidya, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 67340
Record Dates: First submitted 2021-11-17; First posted 2021-12-15 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Catheterization
Keywords: Internal jugular vein; Inferior vena cava; Right heart catheterization
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Right heart catheterization
  Interventions: Device: Ultrasound imaging

INTERVENTIONS:
Device: Ultrasound imaging — Patients scheduled to undergo right heart catheterization (RHC) as their standard of care will be included in the study.
  The patient will be positioned supine at 0 degrees with normal restful breathing and patient looking straight up. After the right sternocleidomastoid muscle is identified, internal jugular vein (IJV) will be imaged at the apex of the triangle formed by the sternal and clavicular heads of the muscle. Similarly, the inferior vena cava (IVC) will be imaged at the caudal end of the sternum. The diameters of both the veins will be noted during normal respiration. The patients will then be asked to sniff and collapsibility of the veins will be noted. No pressure will be applied on the neck. The anticipated duration for image acquisition is between 5 to 10 minutes.
  The patients will undergo the scheduled RHC within 1 hour as scheduled.

SUMMARY:
The study aims to standardize patient positioning during bedside ultrasound assessment of internal jugular vein (IJV) and correlate the results with invasive hemodynamics obtained immediately after. The study hypothesizes that the respiratory variation in the size of IJV, as estimated through ultrasound at bedside, is an accurate estimation of the patient's actual right atrial pressure estimated through right heart catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing right heart catheterization

Exclusion Criteria:

* Superior vena cava obstruction or compression
* Severe tricuspid regurgitation
* Mechanically ventilated patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients scheduled to undergo right heart catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Cross-sectional diameters of the internal jugular vein (IJV) | 5 minutes
  The respiratory variation percentage will assessed using M-mode of the ultrasound while the patient is breathing normally. The maximum and minimum anteroposterior diameter will be noted using M-mode (in mm).
Cross-sectional diameters of the internal jugular vein (IJV) | 5 minutes
  Diameter variation index will be calculated as: (maximum diameter - minimum diameter)/ body surface area.
Sniff collapsibility of IJV | 10 minutes
  Complete collapse (0cm) of the anteroposterior diameter of IJV on sniff maneuver by the patient, as assessed by M-mode on the ultrasound.
Cross-sectional diameters of the inferior vena cava (IVC) | 5 minutes
  Maximum diameter - noted using M-mode (in mm) of the ultrasound machine.
Cross-sectional diameters of the inferior vena cava (IVC) | 5 minutes
  Respiratory variation - assessed using M-mode of the ultrasound while the patient is breathing normally. This will be calculated as (maximum diameter - minimum diameter)/maximum diameter and expressed as a percentage. The maximum and minimum diameters will be noted using M-mode (in mm).
Cross-sectional diameters of the inferior vena cava (IVC) | 5 minutes
  Sniff collapsibility - Complete collapse (0cm) of the cross sectional diameter of IVC on sniff maneuver by the patient, as assessed by M-mode of the ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Gaurang Vaidya, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaidya GN, Kolodziej A, Stoner B, Galaviz JV, Cao X, Heier K, Thompson M, Birks E, Campbell K. Bedside ultrasound of the internal jugular vein to assess fluid status and right ventricular function: The POCUS-JVD study. Am J Emerg Med. 2023 Aug;70:151-156. doi: 10.1016/j.ajem.2023.05.042. Epub 2023 Jun 6. PMID 37307660